CLINICAL TRIAL: NCT04355338
Title: Assessment of Incidence of SARS-CoV-2 Infection and COVID-19 in Brazil
Brief Title: Assessment of Incidence of SARS-CoV-2 Infection and COVID-19 in Brazil (AVISA)
Acronym: AVISA
Status: Completed | Type: Observational
Sponsor: Butantan Institute (Other Government)
Responsible Party: Sponsor
Other Study IDs: COV-01-IB
Record Dates: First submitted 2020-04-17; First posted 2020-04-21 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2024-02

CONDITIONS: COVID-19
Keywords: COVID-19; SARS-CoV-2 infection; Asymptomatic Infections; Antibodies, Neutralizing; Immunity, Humoral
MeSH Terms: conditions — COVID-19; Asymptomatic Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (9):
- 0-9 years: Participants aging 0-9 years
- 10-19 years: Participants aging 10-19 years
- 20-29 years: Participants aging 20-29 years
- 30-39 years: Participants aging 30-39 years
- 40-49 years: Participants aging 40-49 years
- 50-59 years: Participants aging 50-59 years
- 60-69 years: Participants aging 60-69 years
- 70-79 tears: Participants aging 70-79 years
- 80+ years: Participants aging 80 years or more

SUMMARY:
This is an observational study, meaning that no interventions is tested, to determine incidence of SARS-CoV-2 infection and COVID-19 in different clinical sites in Brazil in several age groups. The study aims to assess baseline number of infected participants and perform a follow-up along two years to determine the new cases occurring among participants during the period. All participants will collect blood samples to get more details on the immune response.

DETAILED DESCRIPTION:
This is an observational longitudinal study to assess incidence of SARS-CoV-2 infection in Brazil. The study sample is stratified in nine age groups according decades of life, equally distributed in both sexes, with an expected incidence of 10%, at least, during the study period of 24 months. For the first age groups, (0-9, 10-19 and 20-29 years), sample was calculated with the minimum expected incidence of COVID-19 among infected, regardless severity, is 10%. For the latest age groups (30-39, 40-49, 50-59, 60-69, 70-79 and 80+), the sample was calculated with the expected minimum incidence of hospitalization due to COVID-19 according to estimates per age group reported by Verity R et al. https://doi.org/10.1016/S1473-3099(20)30243-7 After the consent procedure, all participants will have a short interview, a IgG/IgM SARS-CoV-2 rapid test and a blood withdrawal to obtain serum for neutralizing antibodies. These procedures will be repeated every four weeks until the end of the study. Individuals with symptoms compatible will be followed-up to confirm COVID-19 diagnosis as well as to assess severity, need for hospitalization and assisted ventilation, sequels, and eventual reinfection. Levels of neutralizing antibodies and other immune markers will be prospectively assessed in all infected participants, either asymptomatic and symptomatic.

ELIGIBILITY:
Inclusion Criteria:

* Any sex or age
* Providing informed consent
* Agreement with all study visits, procedure and contacts

Exclusion Criteria:

* Previous suspected or confirmed COVID-19
* Febrile illness in the latest 72 hours
* Olfactory or gustatory dysfunction in the last three months
* Healthcare worker in a service with routine attention to COVID-19 patients
* Any conditions that can might hurdle participant's compliance to the study in tha opinion of the study team

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The sample size will be equally distributed in ten different cities of Brazil. Then, each site will have same representation of each age group. Participants can be selected from other ongoing community-based studies conducted in the site and from community in general. Balance of participant according to sex is recommended to the sites in all age group.
Sampling Method: Non-Probability Sample
Enrollment: 3520 (Actual)
Dates: Start 2020-10-25 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Incidence of SARS-CoV-2 infection | 24 months
  Number of cases with serological/virological diagnosis for SARS-Co-2 infection
Incidence of COVID-19 | 24 months
  Number of cases of symptomatic SARS-CoV-2 infection

SECONDARY OUTCOMES:
Incidence of hospitalization due to COVID-19 | 24 years
  Number of cases of hospitalization due to symptomatic SARS-Co-2 infection
Level of neutralizing antibodies | 24 months
  Level of neutralizing antibodies in participants with SARS-Co-2 infection
Previous SARS-CoV-2 infection | 6 months
  Positive serology for SARS-Co-2 infection at baseline

OTHER OUTCOMES:
Incidence of SARS-CoV-2 reinfection | 24 months
  Number of a new SARS-CoV-2 infection in an individual with a proven previous infection
Incidence of COVID-19 cases requiring mechanical ventilation | 24 months
  Number of COVID-19 cases requiring mechanical ventilation
Incidence of deaths due to COVID-19 | 24 months
  Number of deaths due to COVID-19
Incidence of sequels after COVID-19 | 24 months
  Number and description of sequels attributed to COVID-19

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda Boulos, MD, PhD, Study Director — Butantan Institute
Locations (11):
- Brazil (11):
  - Universidade Federal do Ceará, Fortaleza, Ceará
  - Universidade de Brasília, Brasília, Federal District
  - Universidade Federal de Minas Gerais, Belo Horizonte, Minas Gerais
  - Hospital Universitário Júlio Müller da Universidade Federal de Mato Grosso, Cuiabá, Mount
  - Centro de Pesquisas em Medicina Tropical de Rondônia (CEPEM), Porto Velho, Rondônia
  - Universidade Federal de Roraima - UFRR, Boa Vista, Roraima
  - Universidade Federal de Sergipe, Laranjeiras, Sergipe
  - Faculdade de Medicina de São José do Rio Preto - FAMERP, São José do Rio Preto, São Paulo
  - Faculdade Santa Marcelina, São Paulo, São Paulo
  - Hospital Estadual de Serrana, Serrana, São Paulo
  - Instituto de Infectologia Evandro Chagas - Fiocruz, Rio de Janeiro

IPD SHARING:
Plan to Share IPD: No